CLINICAL TRIAL: NCT00176228
Title: Open Trial of Lamotrigine Monotherapy in Pediatric Bipolar Disorder
Brief Title: Lamotrigine Monotherapy in Pediatric Bipolar Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Mani Pavuluri, Professor in Psychiatry, University of Illinois at Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2003-04
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Results first posted 2015-07-30 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2015-06

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Lamotrigine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- lamotrigine (Experimental): The dose of lamotrigine will be 12.5 mg per day beginning the first day. It is increased in 12.5 mg increments every week until it reaches 50 mg and 25 mg per week of increment thereafter until maximum dose of 150 mg in those below 50 kg and 200-400 mg depending on clinical response in those above 50 kg. Increasing the medication to final dose will take 8 weeks and the response on full and tolerable dose is further monitored for response over 6 weeks. Therefore, this is a 18-26 week trial (2 to 12 weeks=screening and wash out; 8 weeks=dosing; 6 weeks=acute trial period on full dose).
  Interventions: Drug: Lamotrigine

INTERVENTIONS:
Drug: Lamotrigine — It is a mood stabilizer that is clinically the first choice if patients present with depression and is effective in adults for mania in maintenance phase. So it is administered to see how effective it is in children and adolescents.
  The dose of lamotrigine will be 12.5 mg per day beginning the first day. It is increased in 12.5 mg increments every week until it reaches 50 mg and 25 mg per week of increment thereafter until maximum dose of 150 mg in those below 50 kg and 200-400 mg depending on clinical response in those above 50 kg.
  Other Names: Lamictal

SUMMARY:
There are two purposes for this project. Study 1 is intended to study the safety and efficacy of Lamotrigine in stabilizing the mood in all phases of pediatric bipolar disorder (Phases: mixed, manic, hypomanic, or depressed episodes) in 8-17 year old children. These children and adolescents must be treatment resistant (who failed on two adequate trials of mood stabilizing medications) to qualify for this study. Study 2 is aimed at examining brain activity and/or dysfunction before lamotrigine treatment, and to look for any alteration after lamotrigine treatment. Brain systems associated with attention and emotional processing will targeted.

DETAILED DESCRIPTION:
Procedure Study 1 This study is planned to be conducted over 18 months, with an average recruitment of 2 subjects per month. Each subject is involved in the study for 18 to 26 weeks. While the study medication is dosed over 8 weeks and treated with full dose over 6 weeks, withdrawal of medications that are on board prior to the study drug administration and drug free period post washout required additional time line that is up to 12 weeks over and above the 14 weeks of administering the study drug. Conversely, the range of time is necessary to account for factors such as the child's age, sex, weight, reactions to the medications and side effects. Based on these factors, the time it takes to titrate the medication dose to the optimal amount will vary. Maintaining this flexibility in the protocol is part of good clinical practice where medication is involved. Only children whose medication is not currently improving their symptoms will be recruited. Therefore no children who have been stabilized on a drug will be taken off of it. The initial 2 week screening period includes a diagnostic interview and collection of demographic information. Previous medication will be tapered slowly over 2-12-week period and is based on tolerability and need to keep subjects in drug free state prior to start of study medication. It is an open trial where subjects are aware of the type of medication and the strength (For example, one pill=25 mg strength) of the pill. Research assessment of mood symptoms and side effects will be carried out 5 times over the course of the active trial period. Blood will be collected 3 times: once the subject is washed-out (baseline), once optimal medication dose has been reached, and finally at the end of the 6-week period on full dose.

The dose of lamotrigine will be 12.5 mg per day beginning the first day. It is increased in 12.5 mg increments every week until it reaches 50 mg and 25 mg per week of increment thereafter until maximum dose of 150 mg in those below 50 kg and 200-400 mg depending on clinical response in those above 50 kg. Increasing the medication to final dose will take 8 weeks and the response on full and tolerable dose is further monitored for response over 6 weeks. Therefore, this is a 18-26 week trial (2 to 12 weeks=screening and wash out; 8 weeks=dosing; 6 weeks=acute trial period on full dose).

Study 2 involves adolescent subjects (>10years of age) recruited from the Study 1 sample. This part of the study is a fMRI treatment study to examine how the brain functions before and after receiving lamotrigine medication for bipolar disorder. The goal of study 2 is to understand how and where lamotrigine works in the brain. In order to do this, we will view brain images in a fMRI scanner pre- and post-treatment. This will be done once before subjects begin taking lamotrigine (subjects who require a "wash-out" period, described in study 1, this will occur after the "wash-out.") The second scan will take place after the medication trial (after the 6-week active treatment period). While in the scanner, subjects will complete tasks related to thinking and emotion. Subjects will be shown pictures of faces with varying expressions including happy, neutral and angry and will be asked to identify the emotions of the faces, remember and identify previously seen faces, and determine the age group of various faces (i.e., above or below 30 years). Subjects will also complete tasks that involve processing words that express different emotions (e.g., happy, angry), and respond to different "go" and "no-go" images that flash on a screen. Brain activity will be recorded during these tasks. Each task will take around 5 minutes. Before the actual fMRI scan, subjects practice lying in a simulator, a machine that looks and sounds like a scanner.

ELIGIBILITY:
Inclusion Criteria:

* Ages 10-20
* Must be able to swallow tablets
* Must be diagnosed with bipolar disorder

Exclusion Criteria:

* Children with general medical condition such as head injury, epilepsy, endocrine disorders
* Those who are on mood altering medications such as steroids, and those diagnosed with mental retardation are excluded to avoid confounding and contributing factors to mood swings.
* If we discover during the interview that the parent and/or child does not understand the consent/assent procedures, we will exclude them.
* Girls who are pregnant or plan to become pregnant during the study period will also be excluded from the research. There have been no concerns raised in the literature about the need for birth control practices in males treated with lamotrigine. As such, there are no provisions to exclude males from the research who do not practice birth control.

We expect only a small number of children to be excluded from the study due to exclusionary criteria. Selection of the subjects is not based on sex, race, or ethnic group.

For the fMRI study:

* Given the limited size of the magnet bore, individuals with a body weight over two-hundred and fifty pounds will be unable to be tested within the MRI scanner.
* Women in the latter stages of pregnancy may be excluded due to large body size and potential discomfort while in the MRI apparatus. Please note that girls who are taking part in the drug portion of the study (this includes all female subjects except the 5 healthy adult, control women) will be given 3 pregnancy during the drug study. This is to rule out pregnancy since pregnant girls should not be taking the study medications for safety reasons.
* Standard contraindications for fMRI studies include: cardiac pacemaker, aneurysm clip, cochlear implants, shrapnel, history of metal fragments in eyes, claustrophobia
* Participants with an IQ of less than 70 (assessed by WRAT) are likely to be excluded due to difficulties comprehending tasks and procedures

Ages: 10 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 48 (Actual)
Dates: Start 2004-02; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mani Pavuluri, MD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- NPI, University of Illinois at Chicago, Chicago, Illinois, United States

REFERENCES:
- [Derived] Pavuluri MN, Passarotti AM, Harral EM, Sweeney JA. Enhanced prefrontal function with pharmacotherapy on a response inhibition task in adolescent bipolar disorder. J Clin Psychiatry. 2010 Nov;71(11):1526-34. doi: 10.4088/JCP.09m05504yel. Epub 2010 Aug 24. PMID 20816040

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In the University of Illinois. The duration of the trial is 14 weeks, with initial 8 weeks of dose titration, followed by 6 weeks of administering the full dose.
Pre-assignment Details: To participate, subjects were required to consent to being washed out of their current medications at study entry. The washout period consisted of tapering their previous medications over one week prior to study entry except for those who received aripiprazole or fluoxetine who required a 4-week washout period.
Groups:
- Lamotrigine: upto 200 mg
Period: Overall Study
Arm/Group | Lamotrigine
Started | 48 (When study began)
Completed | 46 (Study ended)
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Lamotrigine
Number analyzed (Participants) | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 48
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.3 (2.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 21
Region of Enrollment [Number; unit: participants]
  United States | 48

OUTCOME MEASURES:

1. Primary Outcome: Young Mania Rating Scale (YMRS),
Description: This measure has 11 items. The purpose of each item is to rate the severity of that abnormality in the patient. A severity rating is assigned to each of the eleven items, based on the patient's subjective report of his or her condition over the previous forty-eight hours and the clinician's behavioral observations during the interview, with the emphasis on the latter. There are four items that are graded on a 0 to 8 scale (irritability, speech, thought content, and disruptive/aggressive behavior), while the remaining seven items are graded on a 0 to 4 scale. Total score of zero to 60 is possible, zero being normal and 60 being severe, 12 serving as a cut off point for illness if equal or above. There are several ways to show change in outcome. The mean and standard deviation at week 0, 8 and 14 will indicate if there is a change in the scores with the treatment.
Time Frame: Weekly during the 8 week lamotrigine dose titration and 6 week full dose phase.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lamotrigine Effectiveness on YMRS (Mania Measure)
Number analyzed (Participants) | 48
units on a scale
  Baseline | 19.61 (8.94)
  8 week point | 7.06 (6.28)
  14 week point | 5.68 (7.08)

2. Secondary Outcome: Child Depression Rating Scale (CDRS-R)
Description: Response for depressive symptoms was defined as a score less than 40 on the CDRS-R. Range is 18 to 120. Score 18 is normal and higher score signifies depression. The Children's Depression Rating Scale (CDRS) is a 16-item measure used to determine the severity of depression in children 6-18 years of age. Items are measured on 3-, 4-, 5-, and 6-point scales. The mean and standard deviation at week 0, 8 and 14 will indicate if there is a change in the scores with the treatment.
Time Frame: weekly at baseline and each week during osing (8 weeks) and dose stabilized phase (6 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Lamotrigine: Lamotrigine: Response on CDRS-R
Arm/Group | Lamotrigine
Number analyzed (Participants) | 48
units on a scale
  Baseline | 52 (13.25)
  8 week point | 31.39 (12.37)
  14 week point | 26.10 (7.89)

ADVERSE EVENTS:
Arm/Group | Lamotrigine
Serious Adverse Events (participants affected / at risk) | 0/48
Other Adverse Events (participants affected / at risk) | 0/48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No